CLINICAL TRIAL: NCT03058952
Title: Evaluation of a Mindfulness-Based Intervention for Gulf War Illness
Brief Title: Groups for Regaining Our Wellbeing
Acronym: GROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDR 15-197
Record Dates: First submitted 2017-02-07; First posted 2017-02-23 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-02

CONDITIONS: Gulf War; Fatigue; Pain; Depression
Keywords: pain management; fatigue; mindfulness; Gulf War
MeSH Terms: conditions — Fatigue; Pain; Depression; Agnosia | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): An 8-week standardized group program to teach mindfulness skills. In MBSR, participants meet for 2.5 hours per week for 8 weeks in a group format. Participants receive instruction in mindfulness meditation according to a standardized curriculum and have the opportunity to ask questions.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Chronic Disease Self-Management Program (Active Comparator): The CDSMP is a structured program to teach self-management skills based on self-efficacy theory. CDSMP teaches self-management strategies and attempts to modify illness beliefs, enhance self-management capabilities and reinforce successful management strategies. CDSMP is based on self-efficacy theory, which posits that key determinants of behavior are: 1). self-efficacy (confidence in the ability to carry out an action) and 2). outcome expectancy (expectation that a particular goal will be achieved).
  Interventions: Behavioral: Chronic Disease Self-Management Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — An 8-week standardized group program to teach mindfulness skills. In MBSR, participants meet for 2.5 hours per week for 8 weeks in a group format. Participants receive instruction in mindfulness meditation according to a standardized curriculum and have the opportunity to ask questions.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Chronic Disease Self-Management Program — The CDSMP is a structured program to teach self-management skills based on self-efficacy theory. CDSMP teaches self-management strategies and attempts to modify illness beliefs, enhance self-management capabilities and reinforce successful management strategies. CDSMP is based on self-efficacy theory, which posits that key determinants of behavior are: 1). self-efficacy (confidence in the ability to carry out an action) and 2). outcome expectancy (expectation that a particular goal will be achieved).
  Other Names: CDSMP
  Arms: Chronic Disease Self-Management Program

SUMMARY:
This study is a randomized clinical trial measuring outcomes up to 6-months post-intervention. The objective of this study is to evaluate outcomes of two different group interventions for Veterans with Chronic Multisymptom Illness (CMI). The interventions to be compared are Mindfulness-Based Stress Reduction and an adapted version of the Chronic Disease Self-Management Program (aCDSMP) for Veterans experiencing symptoms of Chronic Multi-Symptom Illness (CMI) - musculoskeletal pain, fatigue, and cognitive failures - especially those who were deployed to Gulf War I. Hypothesis One (re: Outcomes): Participants randomized to the adapted Chronic Disease Self-Management Program (aCDSMP) will derive benefit for the primary outcomes, but with smaller effects than the participants randomized to Mindfulness-Based Stress Reduction (MBSR). The investigators hypothesize that Veterans randomized to MBSR will report greater reductions in each of the three primary outcome measures (pain, fatigue, and cognitive failures) at 6-month follow-up as compared to aCDSMP. Hypothesis Two (re: Acceptability): MBSR will be an acceptable and satisfactory program for Veterans with CMI, as measured by attendance rates, a self-report measure of satisfaction, and qualitative interviews. The investigators hypothesize that Veterans with CMI randomized to MBSR will report greater satisfaction with care than their peers randomized to aCDSMP.

DETAILED DESCRIPTION:
The investigators will enroll 308 participants. Half of these will be Gulf War Veterans who meet criteria for CMI, and the other half will be Veterans from other periods of service who also meet criteria for CMI. Each participant will be randomized to either participate in MBSR or aCDSMP (stratified by Gulf War deployment status so there are ~7-8 Gulf War Veterans in each group for every cohort). Measures to collect primary outcome data (pain, fatigue, cognitive failures, patient satisfaction), secondary outcomes, and potential mediators will be administered at four assessments: (1) Baseline; (2) Post-Intervention; (3) at 3-months after the group ended; and (4) at 6-months after the group ended. Sample demographic data (age, gender, race, income, education, etc.) will be collected at baseline only. All study procedures will take place at VA Puget Sound Health Care System in Seattle, WA.

ELIGIBILITY:
Inclusion Criteria:

* Self-report all the criteria for Chronic Multi-Symptom Illness
* Fluent in English and able to provide informed consent

Exclusion Criteria:

* Currently drinking with past-year history of alcohol-related seizures or delirium tremens
* Current DMS-V substance use disorder other than cannabis or nicotine
* Moderate or high risk of suicide as assessed with MINI
* Current psychotic disorder
* Current manic episode
* Diagnosis of borderline personality disorder or antisocial personality disorder
* Inpatient admittance for psychiatric reasons in the past month
* Prior participation in MBSR or CDSMP (attended at least one session)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Simpson, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Only de-identified data, with no individually identifiable patient information, will be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based off of direct mailings generated by a VINCI data pull and the Gulf War Registry, between July 2017 and December 2020. The first participant was enrolled on August 8, 2017, and the last participant was enrolled on December 30, 2020.
Pre-assignment Details: Of 258 enrolled participants, 245 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Started | 123 | 122
Completed Intervention (Completed 6 or more sessions of intervention) | 65 | 65
Completed Immediate Post-assessment | 99 | 96
Completed 3-month Post-intervention Assessment | 97 | 89
Completed | 100 (completed final assessment) | 96 (completed final assessment)
Not Completed | 23 | 26
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 15 | 15
Not completed — Withdrawal by Subject | 7 | 11

BASELINE CHARACTERISTICS:
Population: Note: for the cohort that was receiving intervention that was interrupted by the COVID-19 shutdown in March 2020, 16 participants were removed from the analysis data set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program | Total
Number analyzed (Participants) | 115 | 114 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.4) | 55.6 (8.7) | 56.5 (9.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 14 | 18 | 32
  Gender: Male | 101 | 95 | 196
  Gender: Transgender | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 106 | 103 | 209
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 30 | 23 | 53
  White | 69 | 55 | 124
  More than one race | 3 | 17 | 20
  Unknown or Not Reported | 9 | 12 | 21
Gulf-War Veteran Status [Count of Participants; unit: Participants] — Our definition of Gulf-War Veteran is a Veteran who was deployed to the Gulf War theater of operations any time during August 1990 to August 1991.
  Participants | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Short Form McGill Pain Questionnaire (SF-MPQ-2) Total Score
Description: A validated measure of pain, minimum value: 0, maximum value: 222, higher scores indicate worse outcomes.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on the measure
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 108 | 105
score on scale
  Baseline | 69.2 (42.1) | 64.9 (34.9)
  final 6-month post-intervention: number analyzed (Participants) | 92 | 85
  final 6-month post-intervention | 62.3 (43.4) | 55.5 (38.7)

2. Primary Outcome: General Fatigue Subscale of the Multidimensional Fatigue Inventory (MFI)
Description: A measure of general fatigue symptoms. Minimum value: 0, maximum value: 80, higher scores indicate worse outcomes.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on the measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 114 | 109
score on a scale
  Baseline | 15.1 (3.7) | 14.8 (3.6)
  final 6-month post-intervention: number analyzed (Participants) | 91 | 88
  final 6-month post-intervention | 14.2 (4.1) | 13.6 (4.0)

3. Primary Outcome: Cognitive Failures Questionnaire (CFQ)
Description: A measure of concentration and memory disturbances. Minimum value: 0, maximum value: 100, higher scores indicate worse outcomes.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 111 | 111
score on a scale
  Baseline | 47.0 (18.6) | 49.5 (15.3)
  final 6-month post-intervention: number analyzed (Participants) | 89 | 89
  final 6-month post-intervention | 43.5 (17.3) | 43.5 (14.7)

4. Primary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: A measure of satisfaction with the interventions. Minimum value: 8, maximum value: 32, higher scores indicate higher satisfaction.
Time Frame: report at post-intervention assessment, 3-4 months after baseline
Population: participants who completed at least 1 intervention session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 86 | 83
score on a scale | 25.7 (5.5) | 26.1 (4.6)

5. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: A measure of depression. Minimum value: 0, maximum value: 27, higher scores indicate worse outcomes.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 115 | 114
score on a scale
  Baseline | 9.8 (5.9) | 9.7 (5.9)
  final 6-month post-intervention: number analyzed (Participants) | 92 | 89
  final 6-month post-intervention | 7.8 (6.0) | 7.1 (5.7)

6. Secondary Outcome: PTSD Checklist - Civilian Version (PCL-C)
Description: A measure of PTSD. Minimum value: 0, maximum value: 80. Higher score indicates worse outcome.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on the measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 112 | 112
score on a scale
  Baseline | 31.7 (19) | 31.3 (18.3)
  final 6-month post-intervention: number analyzed (Participants) | 88 | 88
  final 6-month post-intervention | 28.8 (20.5) | 30.3 (18.1)

7. Secondary Outcome: SF-12, Standard (Mental and Physical Component Summary Scores)
Description: A measure of functional status and wellbeing. Two scores generated: a mental component score (MCS) and a physical component score (PCS). For each measure: minimum value: 0, maximum value: 100. Lower score indicates worse outcome.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on the measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 110 | 105
score on a scale
  MCS Baseline | 40.3 (11.5) | 42.3 (11.8)
  MCS final 6-month post-intervention: number analyzed (Participants) | 85 | 81
  MCS final 6-month post-intervention | 43.5 (12.7) | 44.2 (12.4)
  PCS Baseline | 24.7 (8.8) | 23.4 (7.8)
  PCS final 6-month post-intervention: number analyzed (Participants) | 85 | 81
  PCS final 6-month post-intervention | 24.9 (8.8) | 25 (8.3)

8. Secondary Outcome: NIH Patient Reported Outcome Measures Information System (PROMIS) for Alcohol Negative Consequences, Short Form
Description: Substance Use Disorder (SUD) symptom severity for alcohol. Minimum score: 0, maximum score: 35. Higher scores indicate worse outcomes.
Time Frame: Change from baseline to 6 months after completing the intervention
Population: Intent-to-treat population with complete data on the measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
Number analyzed (Participants) | 115 | 114
score on a scale
  Alcohol Negative Consequences Baseline | 4.1 (5.7) | 4.5 (5.5)
  Alcohol Negative Consequences final 6-month post-intervention: number analyzed (Participants) | 90 | 89
  Alcohol Negative Consequences final 6-month post-intervention | 4.7 (6.2) | 5.2 (5.6)

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation, an average of 8-9 months.
Arm/Group | Mindfulness-Based Stress Reduction | Chronic Disease Self-Management Program
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/122
Other Adverse Events (participants affected / at risk) | 2/123 | 0/122
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Stress Reduction (N=123) | Chronic Disease Self-Management Program (N=122)
Hospitalization not due to intervention (Surgical and medical procedures) | 1 (1) | 0 (0) — Veteran was inpatient after multi-symptom organ failure. On ventilator, with palliative care planned.
Suicidal ideation requiring care (Psychiatric disorders) | 1 (1) | 0 (0) — Veteran disclosed thoughts of suicide at post-assessment without plan or intent but in need of immediate care, arranged by research staff

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03058952/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03058952/ICF_001.pdf